CLINICAL TRIAL: NCT01143623
Title: Dose Response Effect of a Proprietary Probiotic Formula for the Prevention of Antibiotic-associated Diarrhea in Chinese Adults
Brief Title: Dose Response Effect of Probiotics for the Prevention of Antibiotic-associated Diarrhea in Chinese Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Cai DongLian, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 09-SBC-2-DAN-03
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Antibiotic-associated Diarrhea
Keywords: antibiotic; diarrhea; probiotic
MeSH Terms: conditions — Diarrhea | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Probiotic (Active Comparator)
  Interventions: Dietary Supplement: Probiotic
- Probiotic-2 (Active Comparator)
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — L. acidophilus, L. paracasei, B. lactis; 2.5 billion cfu capsule once per day
  Arms: Probiotic
Dietary Supplement: Probiotic — L. acidophilus, L. paracasei, B. lactis; 10 billion cfu capsule once per day
  Arms: Probiotic-2
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the dose response effect of probiotic capsules for the prevention of antibiotic-associated diarrhea (AAD).

ELIGIBILITY:
Inclusion Criteria:

* age 30-70 years
* initiating antibiotic therapy
* informed consent

Exclusion Criteria:

* current diarrhea
* life threatening illness
* habitual probiotic use

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Incidence of antibiotic-associated diarrhea | 5 weeks after antibiotic discontinuation

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China